CLINICAL TRIAL: NCT06305858
Title: Partial Versus Total Knee Replacement in Bicompartmental Gonarthrosis (Medial and Patellofemoral): Prospective Functional Assessment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UKA - PFJ
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Knee Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial denture surgical procedure (Experimental)
  Interventions: Procedure: Prosthetic Surgical Procedure
- Total denture surgical procedure with patellar resurfacing (Active Comparator)
  Interventions: Procedure: Prosthetic Surgical Procedure

INTERVENTIONS:
Procedure: Prosthetic Surgical Procedure — The population consists of 48 patients divided into two groups:
  24 patients Group A experimental group: partial denture surgical procedure
  24 patients Group B control group: total denture surgical procedure with patellar resurfacing

SUMMARY:
The study is, in accordance with current legislation, definable as a prospective single-center interventional randomized study.

The aim of the study is to evaluate the post-operative recovery of the group A patient undergoing the partial knee replacement surgical procedure compared to the group B patient undergoing the total knee replacement surgical procedure through clinical/functional scores.

The primary outcome is evaluate the difference in score of the KSS questionnaire, at 1 month after surgery, completed by the patient of group A compared to the patient of group B.

The population consists of 48 adult patients with gonarthrosis divided into two groups:

24 patients Group A experimental group: partial denture surgical procedure

24 patients Group B control group: total denture surgical procedure with patellar resurfacing

DETAILED DESCRIPTION:
The medial unicompartmental prosthesis procedure associated with patellofemoral is reserved for active patients suffering from bicompartmental gonarthrosis in which total knee replacement is to be avoided. The advantage for the patient, compared to total prosthesis surgery, consists in the less invasive nature of the surgical gesture, in the total preservation of the cruciate ligaments and the external compartment and therefore of the native joint biomechanics with the possibility of remote revision with total prosthesis from first implant.

Patients keep "their knee" which is coated and not replaced with advantages in terms of joint feedback and functionality in daily activities and sports practices. This study aims to compare two groups of patients suffering from bicompartmental gonarthrosis (medial and patellofemoral gonarthrosis): Group A undergoing a bicompartmental prosthesis surgical procedure; Group B undergoing a total denture surgical procedure with patellar resurfacing. The two groups will be evaluated with clinical and functional scores aimed at evaluating the outcome in the two surgical procedures.

The number and type of exams are as follows:

* Randomization to Group A or Group B (ad hoc)
* Knee replacement surgery (as usual)
* Compilation of KSS questionnaire at 1, 2, 6, 12 months of follow-up with clinical and functional scores (as a matter of practice)
* Questionnaires and scales (WOMAC, Tegner, VAS and patient satisfaction) at 2, 6, 12 months post intervention (as a matter of practice)
* Recording of any adverse events at 1, 2, 6, 12 months after surgery (as a matter of practice)

ELIGIBILITY:
Inclusion Criteria:

* Grade 3-4 sec Kellgren-Lawrence medial gonarthrosis
* Patellar symptoms
* Primary gonarthrosis
* Patients with ligament integrity
* Age between 40 and 85 years inclusive
* Signing of the Informed Consent and consent to cooperate in all study procedures.

Exclusion Criteria:

* Cognitive impairment
* Psychiatric disorders
* Neuromuscular disorders
* Age > 85 years and <40 years
* Lateral gonarthrosis grade 4 sec Kellgren-Lawrence
* Secondary medial gonarthrosis
* Revisions
* Minors
* Pregnant women self-declaration

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess the difference in score of the KSS (Knee Society Score) questionnaire, completed by the patient in group A compared to the patient in group B | 1 month after surgery
  Evaluate the difference in score of the KSS questionnaire, at 1 month after surgery, completed by the patient of group A compared to the patient of group B

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico San Siro, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided